CLINICAL TRIAL: NCT02235610
Title: Clinical Trial of Ex Vivo Lung Perfusion (EVLP) for the Reconditioning of Marginal Donor Lungs for Transplantation.
Brief Title: Use of Ex Vivo Lung Perfusion (EVLP) in Reconditioning Marginal Donor Lungs for Transplantation
Acronym: EVLP-CHUM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Fondation Pour La Recherche en Chirurgie Thoracique De Montreal (Unknown); Centre de Recherche du Centre Hospitalier de l'Université de Montréal (Other); Institut de Recherches Cliniques de Montreal (IRCM) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CE14.100
Record Dates: First submitted 2014-08-25; First posted 2014-09-10 (Estimated); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Lung Transplant
Keywords: Lung Transplantation; Ex Vivo Lung Perfusion; EVLP

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Group (No Intervention): Recipients receive standard donor lungs as per current clinical practice.
  No experimental procedures will be carried out.
- EVLP Group (Experimental): Recipients receive reconditioned EVLP donor lungs and current standard of care for lung transplant is administered.
  Interventions: Procedure: EVLP Group

INTERVENTIONS:
Procedure: EVLP Group — EVLP technique (Lund Protocol): open left atrium, Steen solution mixed with red blood cells and perfusion 100% of the donor predicted cardiac output.
  Lungs with good and stable function during EVLP will be transplanted into recipients as per current clinical practice.
  Arms: EVLP Group

SUMMARY:
The overall objective of this study is to evaluate the clinical effectiveness of the novel technique of donor EVLP in increasing lung transplant activity by allowing previously unusable donor lungs to be safely used in clinical lung transplantation. Furthermore, to utilize the EVLP technique in research settings thus allowing the evaluation of inflammatory molecules (biomarkers) that would benefit a successful pre-conditioning and increase knowledge of the lungs inflammatory response before transplantation.

DETAILED DESCRIPTION:
Human donor lungs that do not meet the standard clinical criteria for donor lung utilization but fit into the study inclusion criteria will be retrieved from the donor using current donor lung retrieval techniques. These lungs will be brought to the study transplant centre to be perfused in our system by the transplant team. Perfusion of these lungs will be performed using evaluation solution with addition of red blood cells cross matched with the recipient, heparin and antibiotics. Those lungs that after perfusion in our system meet the normal transplantation criteria will be considered for transplantation. Lungs will be excluded for transplantation if the organs don't meet the normal transplantation criteria.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged 18 years and over).
* Patients already on or added to the active waiting list for first lung transplant.
* Patients providing informed consent for participation in the study at the time of study commencement or time of listing for transplant.
* Patients' re-confirmation informed consent for the study on the day of the lung transplant.

Exclusion Criteria:

* Patients aged less than 18 years.
* Patients not providing informed consent for the study.
* Patients not in possession of patient information sheets for the study prior to the day of lung transplant.
* Patients' not re-confirming consent for the study on the day of lung transplant.
* Patients requiring invasive mechanical ventilation, extracorporeal membrane oxygenation (ECMO) support.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-10 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Measure of survival | 12 months after transplantation
  To measure survival 12 months after transplantation in recipients of EVLP assessed and reconditioned donor lungs (treatment group), compared to that of recipients of standard donor lungs (control group), in order to assess whether survival in the EVLP treatment group over that period is non-inferior to that in the standard control group

SECONDARY OUTCOMES:
Evaluate primary graft dysfunction (PGD) | 6h, 12h, 24h, 48h and 72h post-transplant
  PGD is a clinical entity that reflects the development of early acute lung injury after lung transplantation. PGD severity is graded between 0 and 3 and it is measured at 6h, 12h, 24h, 48h and 72 hours after lung transplantation
Duration of hospital stay | Expected average of 6 weeks
  Participants will be followed for the duration of hospital stay, an expected average of 6 weeks
Duration of mechanical ventilation | 30 days after lung transplant
  How long it takes to disconnect the patient from mechanical ventilation
Quality of life (QoL) questionnaire | The day that patients are added to transplant list, at 90 days and 1 year post transplantation
  Questions about Health and Well-Being of patient after lung transplantation
90 day Mortality | 90 days after lung transplant
  Patient survival 90 days after lung transplantation

OTHER OUTCOMES:
Biomarkers | 1 hour pre- and up to 30 days post-transplant
  Measure the concentrations of calgranulin and high mobility group box-1 (HMGB1)

CONTACTS AND LOCATIONS:
Overall Officials: Pasquale Ferraro, MD, Principal Investigator — CHUM
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada